CLINICAL TRIAL: NCT04066725
Title: A Phase II Placebo-controlled Intervention Trial of Oral Aspirin (ASA) as a UV Protectant in Vivo
Brief Title: Aspirin as an Ultraviolet (UV) Protectant in Human Subjects at Risk for Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HCI94424
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Melanoma (Skin)
MeSH Terms: conditions — Melanoma | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ASA 81 mg daily (Experimental): Participants will be given ASA 81 mg orally once daily for a total of 60 days
  Interventions: Drug: Aspirin 81 mg
- ASA 325 mg daily (Experimental): Participants will be given ASA 325 mg orally once daily for a total of 60 days.
  Interventions: Drug: Aspirin 325mg
- Placebo (Placebo Comparator): Participants will be given a placebo orally once daily for a total of 60 days.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Aspirin 81 mg — Participants will be given ASA 81 mg orally once daily for a total of 60 days
  Other Names: ASA
  Arms: ASA 81 mg daily
Drug: Aspirin 325mg — Participants will be given ASA 325 mg orally once daily for a total of 60 days
  Other Names: ASA
  Arms: ASA 325 mg daily
Drug: Placebo oral tablet — Participants will be given placebo orally once daily for a total of 60 days
  Arms: Placebo

SUMMARY:
This is a phase II placebo-controlled intervention trial assessing aspirin (ASA) as a UV protectant in patients at risk for melanoma.

DETAILED DESCRIPTION:
While melanoma risk is largely genetically determined, exposure to ultraviolet (UV) radiation in sunlight is the major environmental risk factor. Although sunscreen use can reduce melanoma risk 2-fold, its efficacy has been questioned, and most patients do not apply sunscreens properly.

This study will evaluate the downstream effects of aspirin (ASA) in human blood and skin moles (nevi) following oral ingestion. We will determine if chronic ingestion of ASA can modulate UV-sensitivity of the skin, UV-induced damage in nevi, and PGE2 levels in blood and nevi.

ELIGIBILITY:
Inclusion Criteria:

* Must have at least 2 nevi (each >5 mm diameter) not clinically suspicious for melanoma that can be biopsied.
* Must be older than age 18.
* Must be able to receive informed consent and sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* The patient cannot speak / understand English or Spanish.
* The patient is pregnant or breastfeeding.
* The patient is a prisoner, critically or mentally ill, or otherwise incapacitated or considered vulnerable.
* The patient has history of allergic reaction to ASA.
* The patient has history of severe asthma.
* The patient has been taking ASA or any NSAID in the past 2 weeks.
* The patient has been taking a blood thinner in the past 2 weeks.
* The patient has history of bleeding disorder.
* The patient has history of peptic ulcer disease.
* The patient has had recent intense UV exposure in the past month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
Change in minimal erythemal dose (MED) from baseline to day 60. | Change from baseline to day 60
  Baseline minimal erythemal dose (MED) measurements will will be compared to MED results at day 60. We will use the conventional definition of MED as the lowest UV dose resulting in erythema that completely fills the 8-mm irradiated site (homogeneous erythema).
Change in concentration of prostaglandin E2 (PGE2) in plasma from baseline to day 60. | Change from baseline to day 60
  Baseline PGE2 levels in plasma specimens will be compared to PGE2 levels at day 60.
Change in concentration of prostaglandin E2 (PGE2) in nevus tissue from baseline to day 60. | Change from baseline to day 60
  Baseline PGE2 levels in tissue specimens will be compared to PGE2 levels at day 60.

SECONDARY OUTCOMES:
Change in concentration of oncometabolite 2-hydroxyglutarate (2-HG) in plasma from baseline to day 60. | Change from baseline to day 60
  Baseline 2-HG levels in plasma specimens will be compared to 2-HG levels at day 60.
Change in concentration of 8-oxoguanine (8-OG) in plasma from baseline to day 60. | Change from baseline to day 60
  Baseline 8-OG levels in plasma specimens will be compared to 8-OG levels at day 60.
Change in concentration of oncometabolite 2-hydroxyglutarate (2-HG) in nevus tissue from baseline to day 60. | Change from baseline to day 60
  Baseline 2-HG levels in tissue specimens will be compared to 2-HG levels at day 60.
Change in concentration of 8-oxoguanine (8-OG) in nevus tissue from baseline to day 60. | Change from baseline to day 60
  Baseline 8-OG levels in tissue specimens will be compared to 8-OG levels at day 60.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Grossman, MD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah, United States